CLINICAL TRIAL: NCT02580877
Title: Exploring Immunologic Effects of Oral Insulin in Relatives at Risk for Type 1
Brief Title: Immune Effects of Oral Insulin in Relatives at Risk for Type 1 Diabetes Mellitus (TN20)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Type 1 Diabetes TrialNet (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Oral Insulin-TN20; UC4DK106993 (NIH); UC4DK117009 (NIH)
Record Dates: First submitted 2015-09-30; First posted 2015-10-20 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Type 1 Diabetes
Keywords: oral insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 67.5 mg oral insulin crystals daily (Experimental): 67.5 mg oral insulin crystals in capsules (by mouth or sprinkled on food) given daily for six months
  Interventions: Drug: 67.5 mg oral insulin crystals daily
- 500mg oral insulin crystals every other week (Experimental): 500 mg oral insulin crystals in capsules (by mouth or sprinkled on food) given every other week for six months
  Interventions: Drug: 500mg oral insulin crystals every other week

INTERVENTIONS:
Drug: 67.5 mg oral insulin crystals daily — human insulin crystals in capsules
  Other Names: Humulin R crystals
  Arms: 67.5 mg oral insulin crystals daily
Drug: 500mg oral insulin crystals every other week — human insulin crystals in capsules
  Other Names: Humulin R crystals
  Arms: 500mg oral insulin crystals every other week

SUMMARY:
The study is a 2 arm, multi-center, randomized, open-labeled clinical trial designed to assess the effects of varying doses and schedules of oral insulin on immunological and metabolic markers in relatives at risk for type 1 diabetes (T1D).

DETAILED DESCRIPTION:
A minimum of 40 eligible participants will be identified for study participation from the TrialNet Pathway to Prevention study. Participants must have a relative with type 1 diabetes and be positive for insulin autoantibodies and at least one other autoantibody. All participants will receive active treatment of recombinant insulin treatment in capsules of either 67.5 mg daily or 500mg every other week. Participants will need to visit the study site up to eleven times over one year for blood tests and other study procedures. During the beginning treatment phase there are two visits one month apart for those given the 67.5 mg dose, and three visits two weeks apart to titrate the dose for those in the 500mg treatment group. There are three additional treatment visits at months 2, 3, and 6 and 4 additional visits for follow-up at months 7, 8, 9 and 12. The primary outcome is the change in immune function as assessed by change in level or quality of T lymphocyte or autoantibody biomarkers measured between 13 and 26 weeks compared to baseline. .

ELIGIBILITY:
Inclusion Criteria:

* Participants in TrialNet Natural History/Pathway to Prevention Study (TN01); is relative of proband with type 1 diabetes
* Between ages 3-45 with normal Oral Glucose Tolerance Test (OGTT) or between ages 3-7 with an abnormal OGTT
* Confirmed positive for insulin autoantibodies within previous six months
* Confirmed positive for one or more other autoantibodies on two separate occasions within the past six months

Exclusion Criteria:

* Diagnosed with type 1 diabetes
* History of treatment with insulin or oral hypoglycemic agent
* History of therapy with immunosuppressive drugs or non-physiologic glucocorticoids within the past two years for a period of more than three months
* Ongoing use of medications known to influence glucose tolerance
* Pregnant or intending to become pregnant while on study or lactating

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2016-01; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Greenbaum, MD, Study Chair — Type 1 Diabetes TrialNet
Locations (19):
- United States (16):
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory Children's Center, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University-Riley Hospital for Children, Indianapolis, Indiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - Columbia University-Naomi Berrie Diabetes Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Benaroya Research Institute, Seattle, Washington
- Walter and Eliza Hall Institute of Medical Research, Parkville, Victoria, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the NIDDK Central Repository
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- [Background] Skyler JS, Krischer JP, Wolfsdorf J, Cowie C, Palmer JP, Greenbaum C, Cuthbertson D, Rafkin-Mervis LE, Chase HP, Leschek E. Effects of oral insulin in relatives of patients with type 1 diabetes: The Diabetes Prevention Trial--Type 1. Diabetes Care. 2005 May;28(5):1068-76. doi: 10.2337/diacare.28.5.1068. PMID 15855569
- [Background] Bonifacio E, Ziegler AG, Klingensmith G, Schober E, Bingley PJ, Rottenkolber M, Theil A, Eugster A, Puff R, Peplow C, Buettner F, Lange K, Hasford J, Achenbach P; Pre-POINT Study Group. Effects of high-dose oral insulin on immune responses in children at high risk for type 1 diabetes: the Pre-POINT randomized clinical trial. JAMA. 2015 Apr 21;313(15):1541-9. doi: 10.1001/jama.2015.2928. PMID 25898052
- [Derived] Jacobsen LM, Schatz DA. Insulin immunotherapy for pretype 1 diabetes. Curr Opin Endocrinol Diabetes Obes. 2021 Aug 1;28(4):390-396. doi: 10.1097/MED.0000000000000648. PMID 34091488

RESULTS

PARTICIPANT FLOW:
Groups:
- 500 mg Oral Insulin Crystals Every Other Week: 500 mg oral insulin crystals in capsules (by mouth or sprinkled on food) given every other week for six months
  500 mg oral insulin crystals every other week: human insulin crystals in capsules
Period: Overall Study
Arm/Group | 67.5 mg Oral Insulin Crystals Daily | 500 mg Oral Insulin Crystals Every Other Week
Started | 45 | 47
Completed | 44 | 43
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 67.5 mg Oral Insulin Crystals Daily | 500mg Oral Insulin Crystals Every Other Week | Total
Number analyzed (Participants) | 45 | 47 | 92
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8.9 [3.8 to 28.1] | 7.9 [3.0 to 43.6] | 8.1 [3.0 to 43.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 25 | 26 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 42 | 41 | 83
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 42 | 42 | 84
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Relationship to person with type 1 diabetes [Count of Participants; unit: Participants]
  Sibling | 34 | 29 | 63
  Parent | 6 | 12 | 18
  Child | 1 | 2 | 3
  Other | 4 | 4 | 8
Glucose Tolerance [Count of Participants; unit: Participants]
  Normal Glucose Tolerance | 36 | 36 | 72
  Abnormal Glucose Tolerance | 9 | 11 | 20
HLA DR3 [Count of Participants; unit: Participants]
  Absent | 31 | 27 | 58
  Present | 14 | 19 | 33
  Unknown | 0 | 1 | 1
HLA DR4 [Count of Participants; unit: Participants]
  Absent | 22 | 15 | 37
  Present | 23 | 31 | 54
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in GAD65 Autoantibody Titer (DK Units/mL)
Description: Change in T-lymphocyte (GAD65) biomarker of beta cell specific immune response
Time Frame: 13 and 26 weeks after first dose versus baseline
Measure: Mean (95% Confidence Interval); unit: DK Units/mL
Arm/Group | 67.5 mg Oral Insulin Crystals Daily | 500 mg Oral Insulin Crystals Every Other Week
Number analyzed (Participants) | 45 | 47
DK Units/mL
  13 weeks | 247 [168 to 363] | 234 [138 to 396]
  26 weeks | 193 [118 to 313] | 196 [121 to 318]

2. Primary Outcome: Change in mIAA Autoantibody Titer From Baseline
Description: Micro-islet autoantibodies (mIAA) autoantibody titers are a measure of of beta cell immune response
Time Frame: 13 and 26 weeks after first dose versus baseline
Measure: Mean (95% Confidence Interval); unit: DK Units/mL
Arm/Group | 67.5 mg Oral Insulin Crystals Daily | 500mg Oral Insulin Crystals Every Other Week
Number analyzed (Participants) | 45 | 47
DK Units/mL
  13 weeks | 0.021 [0.016 to 0.028] | 0.020 [0.015 to 0.028]
  26 weeks | 0.020 [0.015 to 0.028] | 0.017 [0.013 to 0.023]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 1 year
Description: Adverse Events were defined using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Arm/Group | 67.5 mg Oral Insulin Crystals Daily | 500 mg Oral Insulin Crystals Every Other Week
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/47
Other Adverse Events (participants affected / at risk) | 25/45 | 24/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 67.5 mg Oral Insulin Crystals Daily (N=45) | 500 mg Oral Insulin Crystals Every Other Week (N=47)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 4 (5)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Fever (General disorders) | 4 (6) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 4 (5) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (2)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 7 (10) | 2 (2)
Sinusitis (Infections and infestations) | 4 (5) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (7) | 4 (8)
White blood cell decreased (Investigations) | 1 (2) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 3 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT02580877/Prot_SAP_000.pdf